CLINICAL TRIAL: NCT00307567
Title: A Phase II, Multicentre Booster Study to Evaluate Booster Vaccination With GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine or to Evaluate the Immune Memory Following the Administration of a Single Dose of 23-valent Plain Polysaccharide Vaccine in Healthy Children, Previously Vaccinated in Infancy in the Primary Study 11PN-PD-DIT-002 (103488)
Brief Title: Multicentre Booster & Immune Memory Study of a Booster Dose of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine or a Single Dose of 23-valent Plain Polysaccharide Vaccine in Healthy Children Aged 11-18 Mths, Previously Vaccinated in Study 103488
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 105555
Record Dates: First submitted 2006-03-07; First posted 2006-03-28 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Acellular Pertussis; Tetanus; Hepatitis B; Diphtheria; Haemophilus Influenzae Type b; Poliomyelitis
MeSH Terms: conditions — Tetanus; Hepatitis B; Diphtheria; Haemophilus Infections; Poliomyelitis | interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Booster and immune memory study

DETAILED DESCRIPTION:
Total: All 689 subjects enrolled in study 103488. 23PS group: Aventis Pasteurs' 23-valent polysaccharide pneumococcal vaccine (Pneumovax 23) + DTPa-HBV-IPV/Hib; 10V group: GSK Biologicals' 10-valent pneumococcal conjugate vaccine + DTPa-HBV-IPV/Hib

ELIGIBILITY:
Inclusion criteria: Male or female between, and including, 11-18 months of age at the time of vaccination and who previously participated in the study 11PN-PD-DIT-002 and received at least one dose of pneumococcal conjugate vaccine during the primary study, free of obvious health problems and with written informed consent obtained from the parent/guardian of the subject. Exclusion criteria: Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period. Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting one month before the first dose of vaccine(s) and during the entire study period. Administration of any additional pneumococcal vaccine or DTPa combined vaccine since study end of 11PN-PD-DIT-002 study

Ages: 11 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 689
Dates: Start 2005-11; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
1 mth after admin. of booster dose with either GSK Biologicals' 10Pn-PD-DiT vaccine or 1 mth after admin. of single dose of unconjugated 23- valent pneumococcal polysaccharide vaccine (Pneumovax™ 23), anti-pneumococcal serotypes 1,4,5,6B,7F,9V,14,18C,

SECONDARY OUTCOMES:
Pre&post booster: All vaccine pneumococcal serotypes: Opsono titres*
Antibody (Ab) concentrations >= 0.05, 0.20 µg/mL
Ab concentrations to protein D & seropositivity (S+) status
S+/seroprotection status to antigens in DTPa-HBV-IPV/Hib vaccine
Occurrence of: solicited local*,general *symptoms within 4 d
Unsolicited adverse events* within 31 d, SAEs (whole study period) *only post booster

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (43):
- Germany (43):
  - GSK Investigational Site, Bad Saulgau, Baden-Wurttemberg
  - GSK Investigational Site, Bretten, Baden-Wurttemberg
  - GSK Investigational Site, Eppelheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tauberbischofsheim, Baden-Wurttemberg
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Herzogenaurach, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nördlingen, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Koenigstein, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Waren, Mecklenburg-Vorpommern
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Bodenheim, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Schoeneberg - Kuebelberg, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Bredstedt, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Lobenstein, Thuringia
  - GSK Investigational Site, Weimar, Thuringia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 105555 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105555 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105555 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 105555 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105555 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105555 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register